CLINICAL TRIAL: NCT03061968
Title: Study of Appling Acupressure in Low-birth Weight Premature
Brief Title: Study of Applying Acupressure in Low-birth Weight Premature
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Li-Li Chen (Other)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor-Investigator, Li-Li Chen, Principal Investigator, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DMR98-IRB-245-1
Record Dates: First submitted 2011-01-12; First posted 2017-02-23 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Premature
Keywords: acupressure; very-low- birth-weight premature; body weight; behavioral state; developmental status
MeSH Terms: conditions — Premature Birth; Body Weight | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): The babies in experimental group will be observed for one day, and then intervene the simplified acupressure three times a day for fifteen days, and continuously recoding the observation and records until discharge.
  Interventions: Behavioral: acupressure
- control group (No Intervention): The control group only receive routine care in sick baby room unite.

INTERVENTIONS:
Behavioral: acupressure — The babies in experimental group will be observed for one day, and then intervene the simplified acupressure three times a day for fifteen days, and continuously recoding the observation and records until discharge.
  Arms: experimental group

SUMMARY:
The purpose of this study is to investigate the effects of acupressure application in very low birth weight premature.

DETAILED DESCRIPTION:
A quasi-experimental study is designed. Sixty premature babies will be recruited by purposed sampling, according to the criteria of very low birth weight (<1500gm) from a sick baby room in a medical center. The control group only receive routine care in sick baby room unite. The babies in experimental group will be observed for one day, and then intervene the simplified acupressure three times a day for 15 days, and continuously recoding the observation and records until discharge. The intervention includes acupressure for 15 minutes each at 10Am, 1Pm and 4Pm.

ELIGIBILITY:
Inclusion Criteria:

* according to the criteria of very low birth weight (<1500gm) from a sick baby room in a medical center.

Exclusion Criteria:

* Exclusion criteria of very low birth weight (>1500gm) from a sick baby room in a medical center.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 15 days.
  The data will be collected by a self-developed structured questionnaire, including: 1) demographic data of premature; 2)body weight every day until discharge.

IPD SHARING:
Plan to Share IPD: No